CLINICAL TRIAL: NCT06640517
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of Netakimab in Children With Moderate to Severe Plaque Psoriasis
Brief Title: Study of the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of Netakimab in Children With Moderate to Severe Plaque Psoriasis
Acronym: PLANETA-KIDS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-085-16
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — netakimab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NTK (Experimental): netakimab given subcutaneously during main period, open-label period and treatment discontinuation period
  Interventions: Drug: Netakimab
- PBO (Placebo Comparator): placebo given subcutaneously during main period and treatment discontinuation period
  Interventions: Drug: Placebo
- ADA (Active Comparator): adalimumab given subcutaneously during main period
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Netakimab — netakimab will be administered subcutaneously with induction once a week for the first three weeks, then once every 4 weeks
  Arms: NTK
Drug: Placebo — placebo will be administered subcutaneously at a scheme masking netakimab treatment
  Arms: PBO
Drug: Adalimumab — adalimumab will be administered subcutaneously at weeks 1, 2, and then once every 2 weeks
  Arms: ADA

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of netakimab compared with placebo in a pediatric population of subjects over 6 years of age with moderate to severe plaque psoriasis. The study will have randomized, double-blind, placebo-controlled study with open-arm comparison.

DETAILED DESCRIPTION:
Following screening, subjects will be randomized to receive either netakimab, placebo or adalimumab in a 2:1:2 ratio and enter the main study period.

During the main study period, subjects will receive therapy with netakimab/placebo (double-blind arms) or adalimumab (open-label arm), which will be administered subcutaneously until week 12.

At Week 12, after completion of all scheduled procedures subjects in groups netakimab/placebo will continue to receive open-label netakimab for up to week 58, subjects in group adalimumab will switch to open-label adalimumab after 8-week "washout" period.

At Week 58, after completion of all scheduled procedures subjects with sPGA ≤1 will be re-randomised to recieve either netakimab or placebo in double-blind maner. The subjects with >1 will continue to recieve open-label netakimab.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of the legal representative and the subject to participate in the study (the study subject signs the appendix to the information sheet for the legal representative of the clinical study subject with informed consent form).
2. For Stage 1 only: age ≥12 and <18 years at the time of randomization.
3. For Stage 2 only: age ≥6 and <12 years at the time of randomization.
4. A diagnosis of moderate to severe plaque psoriasis with a disease duration of the disease being at least 3 months before the signing of the ICF.
5. Subjects who are candidates for phototherapy or systemic therapy for psoriasis (including non-responders to systemic therapy or phototherapy), in the opinion of the Investigator, or who did not achieve adequate disease control with topical agents.
6. At the time of the screening examination, the body surface area affected by psoriasis is >10% of the body surface area (BSA), the Psoriasis Area and Severity Index (PASI) score is ≥12, and the static Physician's Global Assessment (sPGA) score is ≥3.
7. Subjects with the normal laboratory test results at screening.
8. Subjects with a negative whole blood IFN-γ release test.
9. The ability of the subject and his/her legal representative, in the Investigator's opinion, to perceive information and follow the Protocol procedures.
10. Willingness of subjects and their sexual partners of childbearing potential to use highly effective methods of contraception from the signing of the ICF to 12 weeks after the last dose of the investigational product. This requirement does not apply to subjects who have not reached sexual maturity or who have undergone surgical sterilization. The subject's legal representative must consent to the subject's use of contraception.

Exclusion Criteria:

1. Erythrodermic, pustular, guttate psoriasis, drug-induced psoriasis or any other skin diseases (e.g. eczema) at screening that can affect/complicate the assessment of psoriasis treatment with the investigational product.

2. Use of the following medications:

1. Prior use of drugs based on monoclonal antibodies against interleukin-17 or its receptor.
2. Prior use of adalimumab.
3. Prior use of monoclonal antibodies or their fragments within 12 weeks before signing the ICF.
4. Use of systemic non-biological medicinal products including methotrexate, sulfasalazine, cyclosporine or acitretin within 4 weeks prior to the date of signing the ICF. If previously used systemic non-biologic drugs are discontinued for any reason, the screening period can be extended for up to 8 calendar weeks, during which new systemic non-biologic drugs are not prescribed.
5. Use of phototherapy (including selective phototherapy [UV-B] and photochemotherapy [PUVA]) less than 4 weeks before the date of signing the ICF.
6. Vaccination with live vaccines at any time within 12 weeks prior to signing the ICF or an expected need for such vaccination during the study.

3. Recurrent, chronic, or any other active infection in which, in the opinion of the Investigator, the investigational product may harm the study subject.

4. Sepsis or risk of sepsis. 5. Positive HIV-1 or HIV-2 test. 6. HBV/HCV infections (for details, see Section 6.5.7.2). 7. Established diagnosis or a history of immunodeficiency syndrome (e.g., severe combined immunodeficiency syndrome, T and B cell deficiency syndromes, chronic granulomatous disease), or an infection characteristic of an immunodeficiency (e.g., pneumocystis pneumonia, histoplasmosis or coccidioidomycosis) at the time of signing the ICF.

8. Diagnosis of tuberculosis, including a history of tuberculosis. 9. A clinically significant infection caused by the varicella-zoster virus within 12 weeks prior to signing the ICF.

10. Body temperature ≥38°C at the screening. These subjects may be re-screened, but not earlier than 4 weeks after the first screening.

11. Other concomitant medical conditions that continued at the time of the screening examination, which increase the risk of adverse events during the study or may affect the evaluation of psoriasis symptoms, mask, enhance, or alter the symptoms of psoriasis, or cause clinical or laboratory symptoms similar to those of psoriasis and confirmed by the source documentation:

1. Active inflammatory diseases or aggravation of chronic inflammatory diseases other than psoriasis.
2. Functional class III-IV stable angina of effort, unstable angina or a history of myocardial infarction within 1 year before signing the IC.
3. Moderate to severe cardiac failure (NYHA class III-IV).
4. Grade 2 hypertension.
5. A history of atopic asthma, angioedema.
6. Moderate to severe respiratory failure, Grade 3/4 chronic obstructive pulmonary disease.
7. Decompensated diabetes mellitus; decompensated hypothyroidism, decompensated thyrotoxicosis.
8. Significant systemic autoimmune diseases according to the Investigator.
9. A history of Crohn's disease, ulcerative colitis.
10. Any other underlying conditions (including but not limited to metabolism, hematology, renal, hepatic, pulmonary, neurological, endocrine, cardiac, and gastrointestinal disorders; infections) that may, in the Investigator's opinion, affect the course of psoriasis, affect the assessment of its symptoms, or put the subject using the study therapy at unacceptable risk.

12. Malignant and lymphoproliferative diseases, including lymphoma; symptoms indicating the development of a lymphoproliferative disease (such as lymphadenopathy and/or splenomegaly), except for those previously excluded by a biopsy.

13. History of allergic reactions (anaphylactic shock or allergy to 2 or more drugs).

14. Known allergy or intolerance to monoclonal antibody products or any components of the investigational product.

15. Major surgery within 30 days before the screening, or a major surgery scheduled at any time during the study.

16. Severe infections (including those that required hospitalization or parenteral antibacterial, antimycotic, or antiprotozoal agents) within 6 months prior to signing the ICF.

17. Use of systemic antibacterial, antimycotic, or antiprotozoal agents within 2 months before signing the ICF.

18. More than 4 episodes of respiratory infections over the past 6 months prior to signing the ICF.

19. Any concomitant diseases in which, in the Investigator's opinion, the study therapy may harm the subject.

20. Signs of premature puberty at the screening examination. 21. Pregnancy, breastfeeding, or planning pregnancy while participating in the study.

22. Any psychiatric disorder, including a history of severe depressive disorders and/or suicidal thoughts, which, in the opinion of the Investigator, may pose an excessive risk to the subject or affect the subject's ability to follow the Protocol.

23. Drug addiction, alcoholism, or abuse with drugs or other psychoactive substances (including a history of such disorders).

24. Simultaneous participation in other clinical studies, as well as previous participation in other clinical studies less than 3 months before signing the ICF, prior participation in this study.

25. Use of any other investigational products at the time of signing the ICF or less than 28 days before the planned date of signing the ICF or 5 half-lives (whichever is longer) before the date of signing the ICF.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving PASI75 | Week 12
  PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total body surface area (BSA) affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.
  Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Proportion of subjects achieving sPGA0/1 | Week 12
  Static Physician Global Assessment (sPGA): The physician's global assessment of the Participant's psoriasis lesions at a given time point. Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA assessed as either 0 or 1 represents a clinically meaningful response of minimal plaque severity or complete resolution of plaque psoriasis.

SECONDARY OUTCOMES:
Proportion of subjects achieving PASI75 | Week 58, Week 102
  PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total BSA affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%. Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Proportion of subjects achieving sPGA0/1 | Week 58, Week 102
  Static Physician Global Assessment (sPGA): The physician's global assessment of the Participant's psoriasis lesions at a given time point. Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA assessed as either 0 or 1 represents a clinically meaningful response of minimal plaque severity or complete resolution of plaque psoriasis.
Proportion of subjects achieving IGA mod 2011 0/1 | Week 12, Week 58, Week 102
  Investigator Global Assessment (IGA) mod 2011 provide the assessment of the disease severity from a score of 0 (clear skin) to 4 (severe disease)
Proportion of subjects achieving PASI90 | Week 12, Week 58, Week 102
  PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total BSA affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Proportion of subjects achieving PASI100 | Week 12, Week 58, Week 102
  PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total BSA affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.
  Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Proportion of subjects achieving sPGA0 | Week 12, Week 58, Week 102
  Static Physician Global Assessment (sPGA): The physician's global assessment of the Participant's psoriasis lesions at a given time point. Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA assessed as either 0 or 1 represents a clinically meaningful response of minimal plaque severity or complete resolution of plaque psoriasis.
  An sPGA assessed as 0 represents a clinically important endpoint indicating complete resolution of plaque psoriasis.
Mean change in the PASI score from baseline | Week 12, Week 58, Week 102
  PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total BSA affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.
  Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Mean change in the Nail Psoriasis Severity Index NAPSI from baseline (for subjects with NAPSI>0 at baseline) | Week 12, Week 58, Week 102
  NAPSI is a numeric, reproducible, objective tool for evaluation of nail psoriasis. This scale was used to evaluate the severity of nail bed psoriasis & nail matrix psoriasis by area of involvement in the nail unit. Both fingernail & toenail involvement were assessed.The nail is divided with imaginary horizontal & longitudinal lines into quadrants. Each nail is given a score for nail bed psoriasis (0 to 4) & nail matrix psoriasis (0 to 4), depending on the presence (score of 1) or absence (score of 0) of any of the features of nail bed & nail matrix psoriasis in each quadrant:
  0 = None
  1. = present in one quadrant of nail
  2. = present in two quadrants of nail
  3. = present in three quadrants of nail
  4. = present in four quadrants of nail NAPSI score of a nail is the sum of scores in nail bed & nail matrix from each quadrant (maximum of 8). Each nail is evaluated, & the sum of all the fingernails and toenails is the total NAPSI score ranging from 0 to 160 (No to Severe nail Psoriasis)
Mean change in the pruritus severity score on the numerical rating scale (NRS) from baseline. | Week 12, Week 58, Week 102
  Itch Numeric Rating Scale (NRS): is a single-item, patient-reported outcome (PRO) measure designed to capture the overall severity of a participant's itching due to his/her psoriasis by having the patient circle the integer that describes the worst level of itching in the past 24 hours on an 11-point NRS anchored at 0 representing "no itching" and 10 representing "worst itch imaginable.
Time to relapse defined as sPGA≥2 during the treatment discontinuation period | Week 58 through Week 102
  Static Physician Global Assessment (sPGA): The physician's global assessment of the Participant's psoriasis lesions at a given time point. Plaques are assessed for induration, erythema, and scaling, and an overall rating of psoriasis severity is given using the anchors of clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA assessed as either 0 or 1 represents a clinically meaningful response of minimal plaque severity or complete resolution of plaque psoriasis.
Safety assessment | Through Week 124
  The subjects will be examined for vital signs (blood pressure (BP), wrist pulse rate, axial body temperature) and undergo a physical and instrumental examination, complete blood count, blood chemistry, and urinalysis; the presence and characteristics of adverse events will also be determined. Body weight, height and body mass index will be compared with the World Health Organization's reference values for the physical development of children and adolescents
Immunogenicity assessment | Through Week 102
  Proportion of subjects with detected binding and/or neutralizing antibodies to netakimab.
Pharmacokinetics assessment | Through Week 102
  Multiple dosing pharmacokinetics will be assessed via Ctrough calculation

OTHER OUTCOMES:
Mean change in the PSSI score from baseline (for subjects with PSSI>0 at baseline) | Week 12, Week 58, Week 102
  The scalp is assessed for erythema (redness), induration (hardness), and desquamation (shedding of skin) and percentage of area affected as follows:
  Erythema, Induration and Desquamation:
  0 = Absent
  1. = Slight
  2. = Moderate
  3. = Severe
  4. = Severest Possible
  Percent of Scalp Involved:
  1. <10%
  2. 10% - 29%
  3. 30% - 49%
  4. 50% - 69%
  5. 70% - 89%
  6. 90% - 100% The PSSI score is a composite score derived from the sum of the scores for erythema, induration and desquamation multiplied by the score for the extent of scalp area involved (percent of scalp involved). The range is 0 (no psoriasis) to 72 (Most severe Disease).
Mean change in the PPASI score from baseline (for subjects with PPASI>0 at baseline) | Week 12, Week 58, Week 102
  Both the palms & soles on each hand & foot is assessed for erythema, induration, desquamation & percentage of area affected as follows:
  Erythema (E), Induration (I), & Desquamation (D):0 = None, 1 = Slight, 2 = Moderate, 3 = Severe, 4 = Very Severe
  Percent of Palm and Sole Area Covered:
  0 = None, 1 = <10%, 2 = 10% - 29%, 3 = 30% - 49%, 4 = 50% - 69%, 5 = 70% - 89%, 6 = 90% - 100% PPASI score is a composite score derived from the sum scores for E, I, & D multiplied by a score for the extent of palm & sole area involvement. The range is 0 (no psoriasis) to 72 (most severe disease).
Mean change in the mGPASI score from baseline (for subjects with mGPASI>0 at baseline) | Week 12, Week 58, Week 102
  Genital area is assessed for erythema, induration, desquamation & percentage of area affected as follows:
  Erythema (E), Induration (I), & Desquamation (D):0 = None, 1 = Slight, 2 = Moderate, 3 = Severe, 4 = Very Severe
  Percent of Genital Area Covered:
  0 = None, 1 = <10%, 2 = 10% - 29%, 3 = 30% - 49%, 4 = 50% - 69%, 5 = 70% - 89%, 6 = 90% - 100% mGPASI score is a composite score derived from the sum scores for E, I, & D multiplied by a score for the extent of area involvement. The range is 0 (no psoriasis) to 72 (most severe disease).
Proportion of subjects achieving CDLQI/DLQI0/1 | Week 12, Week 58, Week 102
  DLQI is a validated, dermatology-specific, patient reported measure that evaluates participant's health-related quality of life. It consists of 10 items that are grouped in 6 domains: symptoms & feelings, daily activities, leisure, work & school , personal relationships, & treatment. The recall period of this scale is over the "last week." Response categories and corresponding scores are:
  Very much = 3, A lot = 2, A little = 1, Not at all = 0, Not relevant = 0. A DLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment). CDLQI questionnaire is designed for use in children (4 to 16 years of age). It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. A CDLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment).
Mean change in the CDLQI/DLQI quality of life score from baseline | Week 12, Week 58, Week 102
  DLQI is a validated, dermatology-specific, patient reported measure that evaluates participant's health-related quality of life. It consists of 10 items that are grouped in 6 domains: symptoms & feelings, daily activities, leisure, work & school , personal relationships, & treatment. The recall period of this scale is over the "last week." Response categories and corresponding scores are:
  Very much = 3, A lot = 2, A little = 1, Not at all = 0, Not relevant = 0. A DLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment). CDLQI questionnaire is designed for use in children (4 to 16 years of age). It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. A CDLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment).

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Federal State Budgetary Educational Institution of Higher Education "Altai State Medical University" of the Ministry of Health of the Russian Federation, Barnaul
  - State budgetary healthcare institution "Chelyabinsk Regional Clinical Dermatovenerological Dispensary", Chelyabinsk
  - Limited Liability Company "Health Azbuka Medical Center", Kazan'
  - State Autonomous Healthcare Institution "Republic Clinical Dermatovenerologic Dispensary of the Ministry of Health of the Republic of Tatarstan named after Professor Ge", Kazan'
  - State Autonomous Healthcare Institution "Kuzbass Clinical Dermatovenerological Dispensary", Kemerovo
  - Federal State Budgetary Educational Institution of Higher Education "Kirov State Medical University" of the Ministry of Health of the Russian Federation, Kirov
  - State budgetary healthcare institution "Clinical Dermatovenerologic Dispensary" of the Ministry of Health of the Krasnodar Territory, Krasnodar
  - Federal State Autonomous Institution "National Medical Research Center for Children's Health" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Institution "State scientific centre of dermatovenerology and cosmetology" of the Ministry of health of Russian Federation, Nizhny Novgorod branch, Nizhny Novgorod
  - Federal State Budgetary Educational Institution of Higher Education "St. Petersburg State Pediatric Medical University" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Limited Liability Company "PiterKlinika", Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Siberian State Medical University" of the Ministry of Health of the Russian Federation, Tomsk
  - Federal State Budgetary Educational Institution of Higher Education "Siberian State Medical University", Tomsk
  - State budgetary institution of the Sverdlovsk region "Ural Research Institute of Dermatovenereology and Immunopathology", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No